CLINICAL TRIAL: NCT04952272
Title: Intratumor CpG-ODN Injection Boosters Immune Killing Against in Situ Tumor Antigen Released by Interventional Approaches for Advanced Solid Tumors
Brief Title: Intratumor CpG-ODN Injection Boosters Immune Killing Against in Situ Tumor Antigen Release for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Guangdong Zhaotai InVivo Biomedicine Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZITCpG-013
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Hepatocellular Carcinoma; Solid Tumor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Hepatocellular | interventions — CPG-oligonucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratumor CpG-ODN Injection (Experimental): CpG-ODN will be Injected into the tumor.
  Interventions: Combination Product: CpG-ODN

INTERVENTIONS:
Combination Product: CpG-ODN — CAR-T cells secreting scFv against OX40
  Other Names: Interventional therapy technique including microwave ablation or drug-eluting beads

SUMMARY:
To study the safety and clinical effects of intratumor injecting CpG-ODN and in situ release of tumor antigen by interventional ablation or drug-eluting beads to treat advanced solid tumors.

DETAILED DESCRIPTION:
1. Percutaneous microwave ablation or intratumor injection of drug-eluting beads to destroy cancer cells to release tumor-specific antigens
2. Intratumor injection of type A/C CpG-ODN with or without infusion of CAR-T cells secreting scFv against OX40
3. Assessing side effects and therapeutic efficacy after the combined treatments

ELIGIBILITY:
Inclusion Criteria:

* Solid advanced malignant tumors
* Age between18 and 80 years
* Life expectancy is greater than three months

Exclusion Criteria:

* Benign tumor
* Life expectancy is less than three months
* Serious medical comorbidity
* Others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2036-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessing safety and treatment efficacy on intratumor injection of CpG-ODN and in situ tumor antigen release for advanced tumors | up to 36 months
  Assessing incidence of side effects and primary clinical response of the intratumor injection of CpG-ODN and therpeutical in situ tumor antigen release for advanced tumors, including CR, PR, SD, and PD.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No